CLINICAL TRIAL: NCT01693887
Title: A Comparative Study About Empirical Therapy and Preemptive Therapy to Invasive Pulmonary Fungal Infection ICU Patients in China
Brief Title: Treatment Method Research of Invasive Pulmonary Fungal Infection
Acronym: 4056
Status: Terminated | Type: Observational
Why Stopped: The study difficulty is more serious than expected. The budget isn't enough.
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, yan kang, director（ICU）, West China Hospital
Other Study IDs: ITRFUN4056
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: IFI
Keywords: IFI; empirical therapy; preemptive therapy; Itraconazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- empirical therapy: immediate initiation of antifungal therapy; Itraconazole :1-14day,iv；(400mg/day bid 1-2day, 200mg/day q.d 3-14day) 15-28day,p.o(400mg/day bid)
- preemptive therapy: Dynamic monitoring of fungal infection, initiation antifungal therapy when clinical diagnosis ( microbial + experiment +, G/GM, CT typical change ) approveled in two weeks Itraconazole :1-14day,iv；(400mg/day bid 1-2day, 200mg/day q.d 3-14day) 15-28day,p.o(400mg/day bid) If within two weeks without obtaining positive results, researchers determine whether initiation of antifungal therapy。

SUMMARY:
The purpose of this study is to Comparison clinical efficiency with IPFI patients who treated by different protocols(empirical therapy or preemptive therapy) in ICU.

DETAILED DESCRIPTION:
a multicenter study ( a total of 2411 person-time ) found In the United States in 205, antifungal therapy in empirical therapy, preemptive therapy, target therapy of respectively 44%, 43%, 12%. While the existing on preemptive therapy and empiric treatment comparative study shows, the survival rate of the patients without differences, cost and application of antifungal drugs are relatively more in empirical therapy. These findings of differences, is due to the different research forecast model, treatment options vary widely, and are without a prospective multicenter study of verification. Initiation of antifungal therapy time and antifungal drug of choice is affected by many factors, including the risk stratification of patients, clinical manifestations, bacterial infection of evidence and non interventional diagnosis method results. How to grasp the opportunity to treat the fungal infections by empirical therapy or preemptive therapy that has plagued the global clinical doctors. The purpose of this study is aimed at the large scale prospective, multicenter study method to China, severe invasive pulmonary fungal infection of the empiric treatment with preemptive therapy for clinical contrast research, exploration of fungal treatment time and plan, to establish China's own optimal antifungal treatment options, are reduced in patients with severe fungal infection harm and increase the rate of successful treatment with evidence-based medical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old ，male or female
2. Expected the time of staying in ICU longer than 72 hours and the duration of mechanical ventilation for more than 48 hours
3. Pulmonary infection according to, axillary temperature≥ 37℃, using broad-spectrum antibiotics more than 72 hours, no better or worse
4. Candida score greater than or equal to 3
5. Child-bearing women, urine pregnancy test must be negative when screening and agreed to adopt safe and effective contraceptive measures in the process
6. Male subjects must be guaranteed to use dual physical methods of contraception contraceptive and sperm donation, from starting to after 30days ending treatment
7. Subjects ( or their legal representatives） have signed the informed consent

Exclusion Criteria:

1. Diagnosed with invasive fungal infection by any of the following means at the time of admission 1）Proved deep fungal infection by histopathology 2）Peripheral blood culture fungi positive at least 1 time 3）Specimens from sterile sites of culture positive ( cerebrospinal fluid, pleural effusion and ascites）
2. Renal insufficiency, creatinine clearance < 30ml/min
3. Active liver disease or suspected drug induced liver injury
4. Pregnant and lactating women
5. With imidazole or pyrrolic drug allergy or intolerance or have contraindications.
6. Not fit into the group by comprehensive judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: suspected Pulmonary invasive fungal Infection in ICU patients with Mechanical Ventilation
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: yan kang, director, Principal Investigator — West China Hospital; xiao bo huang, director, Study Director — Sichuan Provincial People's Hospital; chuan zhang, director, Study Director — Third people's Hospital of Chengdu City; di-fen wang, director, Study Director — Affiliated Hospital of Guiyang Medical College
Locations (4):
- China (4):
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - Third people's Hospital of Chengdu City, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - Sichuan provincial people's hospital, Chengdu, Sichuan